CLINICAL TRIAL: NCT06494774
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses and Multiple Oral Doses Over 10 Days of BI 1815368 in Japanese Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Different Doses of BI 1815368 Are Tolerated and How BI 1815368 is Taken up in the Body of Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1485-0005
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SRD part: low dose (Experimental): Single-rising dose (SRD)
  Interventions: Drug: BI 1815368
- SRD part: medium dose followed by MD part (Experimental): Single-rising dose (SRD) Multiple dose (MD)
  Interventions: Drug: BI 1815368
- SRD part: high dose (Experimental)
  Interventions: Drug: BI 1815368
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1815368

INTERVENTIONS:
Drug: BI 1815368 — BI 1815368
  Arms: SRD part: high dose; SRD part: low dose; SRD part: medium dose followed by MD part
Drug: Placebo matching BI 1815368 — Placebo matching BI 1815368
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability. pharmacokinetics (PK), and pharmacodynamics of BI 1815368 in healthy Japanese male subjects following administration of single rising doses or multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12- lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 25 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Japanese ethnicity, according to the following criteria: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 40 to 90 mmHg, or pulse rate outside the range of 40 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | Up to 26 days

SECONDARY OUTCOMES:
SRD part: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 6 days
  Single-rising dose (SRD)
SRD part: Maximum measured concentration of the analyte in plasma (Cmax) | Up to 6 days
  Single-rising dose (SRD)
MD part: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to 19 days
  Multiple dose (MD)
MD part: Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Up to 19 days
  Multiple dose (MD)
MD part: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Up to 19 days
  Multiple dose (MD)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com